CLINICAL TRIAL: NCT00817063
Title: Efficacy and Safety of Alitretinoin in the Treatment of Severe Chronic Hand Eczema Refractory to Topical Therapy
Brief Title: Efficacy and Safety of a Retinoid in the Treatment of Severe Chronic Hand Eczema
Acronym: HANDEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 117183; BAP01346 (Other: Basilea Pharmaceutica); NCT00817063 (Registry Identifier: Clinicaltrials.gov)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Eczema
Keywords: retinoid treatment; fingertip dermatitis; hyperkeratotic hand eczema; vesicular hand eczema; pompholyx
MeSH Terms: conditions — Eczema; Eczema, Dyshidrotic | interventions — Alitretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alitretinoin (Experimental): Patients will receive alitretinoin 30mg capsule for up to 24 weeks
  Interventions: Drug: alitretinoin
- Placebo (Experimental): Patients will receive placebo 30mg capsule for up to 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alitretinoin — Patients receive alitretinoin 30mg one capsule daily for up to 24 weeks
  Arms: Alitretinoin
Drug: Placebo — Patients receive matching placebo for up to 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of alitretinoin in the treatment of severe chronic hand eczema that does not respond to treatment with potent topical steroids.

DETAILED DESCRIPTION:
Chronic hand eczema (CHE)is a distressing disease that poses difficult problems for dermatologists. CHE leads to considerable work-absenteeism, disability and exclusion from labour market. Conventional treatments, including highly potent topical steroids, yield often unsatisfactory results. This study investigates the efficacy and safety of oral alitretinoin, a retinoid, in patients who have not responded to avoidance of causative factors, such as contact allergens and skin irritants, non-medicated skin care and highly potent topical steroids. Eligible patients are randomly assigned to receive alitretinoin or a placebo.

ELIGIBILITY:
Inclusion Criteria:

* all types of chronic hand eczema, lasting for at least 6 months since initial diagnosis
* rated as severe by the physician
* unresponsive to highly potent topical corticosteroids, such as clobetasol

Exclusion Criteria:

* patients whose disease is adequately controlled by standard non-medicated therapy, including potent topical steroids, skin moisturizers, and avoidance of allergens and irritants
* patients with known allergens and irritants, who have not made a reasonable effort to avoid the substances
* patients with psoriasis lesions
* active fungal, bacterial or viral infections of the hands
* female patients who are pregnant or breastfeeding
* female patients of childbearing potential who cannot use or will not commit to use two effective methods of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2009-01-08 (Actual); Primary Completion 2012-04-26 (Actual); Study Completion 2012-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (70):
- United States (70):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Radiant Research Inc., Tucson, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Hull Dermatology, Rogers, Arkansas
  - Shahram Jacobs, MD, Inc., Encino, California
  - University of California, San Diego Dermatology Clinical Trials Unit, La Jolla, California
  - Dermatology Research Associates, Los Angeles, California
  - Laser and Dermatology Center, Marina del Rey, California
  - Integrated Research Group, Riverside, California
  - University of California, Davis, Sacramento, California
  - Therapeutics Clinical Research, San Diego, California
  - East Bay Psoriasis Treatment Center, San Ramon, California
  - Stanford University Dept of Dermatology, Stanford, California
  - Solano Clinical Research, Dow Pharmaceutical Sciences, Vallejo, California
  - Longmont Clinic, P.C., Longmont, Colorado
  - Western State Clinical Research Inc., Wheat Ridge, Colorado
  - George Washington University - Medical Faculty Associates, Washington D.C., District of Columbia
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Toccoa Clinic Medical Associates, Toccoa, Georgia
  - Saltzer Medical Group, Nampa, Idaho
  - Michael Bukhalo MD, Arlington Heights, Illinois
  - Dermassociates, Ltd, Belleville, Illinois
  - Schaumburg Dermatology, Schaumburg, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Indiana University Dermatology, Indianapolis, Indiana
  - The Dermatology Center, New Albany, Indiana
  - Dermatology Center of Indiana/Indiana Clinical Trials Center, Plainfield, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - American Dermatology Association, Shawnee Mission, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Dermatology Specialists, Louisville, Kentucky
  - Derm Research, PLLC, Louisville, Kentucky
  - Tulane University Health Sciences, Dermatology Dept, New Orleans, Louisiana
  - Hamzavi Dermatology Clinic, Fort Gratiot, Michigan
  - Silverton Skin Institute, Grand Blanc, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - MAPS Applied Research Center, Edina, Minnesota
  - Minnesota Clinical Studies Research Center, Fridley, Minnesota
  - Washington University Dermatology Research, St Louis, Missouri
  - South Lincoln Dermatology, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - UMDNJ - Robert Wood Johnson School of Medicine, Dermatology, Somerset, New Jersey
  - St.Luke's/Roosevelt Hospital Center, New York, New York
  - Mount Sinai School of Medicine Clinical Dermatology, New York, New York
  - Helendale Dermatology and Medical Spa, Rochester, New York
  - Derm Research Center of New York Inc., Stony Brook, New York
  - University of North Carolina, Dermatology Department, Chapel Hill, North Carolina
  - Azalea Research Center, Wilmington, North Carolina
  - Wake Forrest University School of Medicine, Winston-Salem, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Paddington Testing Co.Inc, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Dermatology Associates of Kingsport, Kingsport, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Academy of Clinical Research, Arlington, Texas
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Virginia Clinical Research Inc., Norfolk, Virginia
  - Dermatology and Laser Center NW, Bellingham, Washington
  - Premier Clinical Research, Seattle, Washington
  - Madison Skin & Research Inc., Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD for this study will be made available via the Clinical Study Data Request site.
Access Criteria: IPD for this study will be made available via the Clinical Study Data Request site.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20099

REFERENCES:
- [Background] Diepgen TL, Agner T, Aberer W, Berth-Jones J, Cambazard F, Elsner P, McFadden J, Coenraads PJ. Management of chronic hand eczema. Contact Dermatitis. 2007 Oct;57(4):203-10. doi: 10.1111/j.1600-0536.2007.01179.x. PMID 17868211
- [Background] Ruzicka T, Larsen FG, Galewicz D, Horvath A, Coenraads PJ, Thestrup-Pedersen K, Ortonne JP, Zouboulis CC, Harsch M, Brown TC, Zultak M. Oral alitretinoin (9-cis-retinoic acid) therapy for chronic hand dermatitis in patients refractory to standard therapy: results of a randomized, double-blind, placebo-controlled, multicenter trial. Arch Dermatol. 2004 Dec;140(12):1453-9. doi: 10.1001/archderm.140.12.1453. PMID 15611422
- [Background] Ruzicka T, Lynde CW, Jemec GB, Diepgen T, Berth-Jones J, Coenraads PJ, Kaszuba A, Bissonnette R, Varjonen E, Hollo P, Cambazard F, Lahfa M, Elsner P, Nyberg F, Svensson A, Brown TC, Harsch M, Maares J. Efficacy and safety of oral alitretinoin (9-cis retinoic acid) in patients with severe chronic hand eczema refractory to topical corticosteroids: results of a randomized, double-blind, placebo-controlled, multicentre trial. Br J Dermatol. 2008 Apr;158(4):808-17. doi: 10.1111/j.1365-2133.2008.08487.x. Epub 2008 Feb 21. PMID 18294310
- [Derived] Fowler JF, Graff O, Hamedani AG. A phase 3, randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of alitretinoin (BAL4079) in the treatment of severe chronic hand eczema refractory to potent topical corticosteroid therapy. J Drugs Dermatol. 2014 Oct;13(10):1198-204. PMID 25607554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 599 participants were randomized, out of these 3 participants did not receive study medication, hence Intent-to-treat (ITT) population consisted of 596 participants which included all randomized participants who were dispensed medication.
Pre-assignment Details: A total of 942 participants entered the run-in period for a maximum of 16 weeks who received class 1 corticosteroids for 2 weeks followed by corticosteroids of any potency. Out of 942 participants, 343 participants were run-in failures and hence 599 were randomized in the study.
Groups:
- Alitretinoin 30 mg: Participants with severe CHE rated as refractory during the run-in period were randomized to receive 30 milligrams (mg) of alitretinoin oral soft capsule once daily up to 24 weeks.
- Placebo: Participants with severe CHE rated as refractory during the run-in period were randomized to receive matching Placebo oral soft capsule once daily up to 24 weeks.
Period: Overall Study
Arm/Group | Alitretinoin 30 mg | Placebo
Started | 298 | 298
Completed | 161 | 128
Not Completed | 137 | 170
Not completed — Adverse Event | 32 | 13
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 33 | 86
Not completed — Failure to Return | 13 | 12
Not completed — Violation of Selection at Entry | 7 | 4
Not completed — Protocol Violation | 3 | 8
Not completed — Withdrawal by Subject | 17 | 37
Not completed — Early Improvement | 19 | 4
Not completed — Administrative | 10 | 4
Not completed — Abnormality of Laboratory Test | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Alitretinoin 30 mg: Participants with severe CHE rated as refractory during the run-in period were randomized to receive 30 mg of alitretinoin oral soft capsule once daily up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Alitretinoin 30 mg | Placebo | Total
Number analyzed (Participants) | 298 | 298 | 596
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (12.55) | 47.5 (12.96) | 47.3 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 149 | 282
  Male | 165 | 149 | 314
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 15 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 35 | 54
  White | 263 | 238 | 501
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Responded as Per Physician's Global Assessment (PGA) at Week 24
Description: The investigator assigned PGA grades according to a 5-point scale (clear [not detectable], almost clear [less than 10% of affected hand surface], mild disease [less than 10% of affected hand surface], moderate disease [10% to 30% of affected hand surface], severe disease [>30% of affected hand surface]). PGA ratings were based on an integrated clinical picture of signs, symptoms, and the extent of disease. Symptoms included erythema, scaling, hyperkeratosis/lichenification, vesiculation, edema, fissures, and pruritus/pain. The PGA scale ranges from 0 (no symptom) to 4 (severe disease). Participants were considered as responders when they had a PGA of clear or almost clear.
Time Frame: Week 24 (end-of-treatment)
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 298 | 298
Participants
  Clear | 58 | 14
  Almost clear | 60 | 30
  Total | 118 | 44
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Odds Ratio (OR) = 3.78, 95% CI 2-sided [2.55 to 5.62]
Statistical Analysis 2: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Difference in Percentage = 24.8, 95% CI 2-sided [18.0 to 31.7]

2. Secondary Outcome: Percentage Change From Baseline in Modified Total Lesion Symptom Score (mTLSS) at the End-of-treatment
Description: A 4-point scale (0=none, 1=mild, 2=moderate, 3=severe) was used to grade 7 signs or symptoms of CHE. The mTLSS was calculated as sum of assigned scores for the symptoms of erythema, scaling, lichenification/hyperkeratosis, vesiculation, edema, fissures and Pruritus/Pain. The total score ranged from 0 (best) to 21 (worst). Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-baseline values. Percentage change from Baseline = (change from Baseline / Baseline value) * 100. Data for Week 24 last observation carried forward (LOCF) has been presented.
Time Frame: Baseline (Week 0) and Week 24 (end-of-treatment)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 298 | 298
Percent change | -53.99 (40.160) | -29.86 (37.830)
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p < 0.001, Kruskal-Wallis; Mean Difference (Net) = -24.13, 95% CI 2-sided [-30.40 to -17.85]

3. Secondary Outcome: Number of Participants Who Responded as Per Patient Global Assessment (PaGA) at End-of-treatment
Description: At Week 24 or at the end-of-treatment participants were asked by the investigator to grade their overall change from Baseline by selecting one of the following descriptions, which best matched their perception of overall treatment effect: cleared or almost cleared (at least 90% clearing), marked improvement (at least 75% clearing), moderate improvement (at least 50% clearing), mild improvement (at least 25% clearing), no change and worsening. Participants were considered as responders when the PaGa was cleared or almost cleared.
Time Frame: Week 24 (end-of-treatment)
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 298 | 298
Participants | 117 | 41
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Odds Ratio (OR) = 4.05, 95% CI 2-sided [2.71 to 6.07]
Statistical Analysis 2: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Difference in Percentage = 25.5, 95% CI 2-sided [18.7 to 32.3]

4. Secondary Outcome: Percentage Change From Baseline in Extent of Disease at End-of-treatment
Description: The extent of disease was estimated as the percentage of hand area (with 100% defined as the palmar and dorsal aspects) affected by eczema at Baseline, and at the end of treatment). Extent of disease was estimated separately for the left and right hands, and the overall extent of disease for both hands was calculated as (Left+Right)/2. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-baseline values. Percentage change from Baseline = (change from Baseline / Baseline value) * 100.
Time Frame: Baseline (Week 0) and Week 24 (end-of-treatment)
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 271 | 269
Percent change | -46.56 (53.746) | -24.20 (48.214)
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p < 0.001, Kruskal-Wallis; Mean Difference (Net) = -22.36, 95% CI 2-sided [-31.00 to -13.73]

5. Secondary Outcome: Response Duration for Responding Participants at the End-of-therapy
Description: Response Duration was defined as time from the end-of-therapy to the first diagnosis of mild, moderate, or severe CHE. Median and inter-quartile range has been presented.
Time Frame: Up to 72 Weeks (including 24 weeks of treatment and 48 weeks of follow-up)
Population: ITT population.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 298 | 298
Weeks | 8.3 [4.7 to 16.7] | 16.9 [5.1 to 50.3]
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p = 0.047, Log Rank

6. Secondary Outcome: Time to Relapse for Responding Participants at the End-of-therapy
Description: Time to relapse was defined as the time from end-of-therapy to the first diagnosis of severe CHE. Median and inter-quartile range has been presented. The median was based on the very last participant having a follow-up period longer than expected, those explaining the high median.
Time Frame: Up to 72 Weeks (including 24 weeks of treatment and 48 weeks of follow-up)
Population: ITT population.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 298 | 298
Weeks | 83.0 [18.1 to 83.0] | NA [39.6 to NA] — An analysis of the time to relapse from the End-of-therapy did not have sufficient data to yield a good estimate of median time to relapse as well as for Q3.
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p = 0.068, Log Rank

7. Secondary Outcome: Time to Response for Responding Participants at End-of-therapy
Description: Time to response was defined as time from start of treatment to first PGA assessment of "clear" or "almost clear". Median and inter-quartile range has been presented.
Time Frame: Up to 72 Weeks (including 24 weeks of treatment and 48 weeks of follow-up)
Population: ITT population. Only those participant who responded to PGA assessment at the end of therapy was analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 118 | 44
Days | 65.0 [54.0 to 112.0] | 117.0 [85.0 to 167.0]
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Test type: Superiority; p < 0.001, Log Rank

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Treatment Period
Description: An AE was defined as any adverse change from the participant's Baseline (pretreatment) clinical condition, including intercurrent illness, which occurred during the course of the clinical study after written informed consent had been given, whether considered related to treatment or not. A treatment-emergent AE was defined as any adverse change that occurred after treatment started and up to 7 days after last treatment. An SAE was any experience that suggested a significant hazard, contradiction, side effect or precaution. It was any adverse event that at any dose resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect.
Time Frame: Up to Week 24 (end-of-treatment)
Population: Safety Population included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Participants
  Any AEs | 216 | 155
  Any SAEs | 7 | 3

9. Secondary Outcome: Number of Participants With Maximum Post Baseline Laboratory Values Outside the Marked Reference Range
Description: Blood samples were collected for the assessment of laboratory parameters hemoglobin, hematocrit, erythrocytes, mean corpuscular volume, mean corpuscular hemoglobin concentration, reticulocytes, platelets, white blood cell, lymphocytes, neutrophils, monocytes, eosinophils, basophils, total bilirubin, bilirubin conjugated (direct), aspartate amino transferase (AST), alanine amino transferase (ALT), lactate dehydrogenase (LDH), creatine phosphokinase (CPK), alkaline phosphatase (ALP), total protein, serum albumin, glucose, triglycerides, total cholesterol, high-density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, sodium, potassium, chloride, serum calcium, serum phosphate, serum creatinine, blood urea nitrogen (BUN)/urea, uric acid, Free thyroxin and thyroid stimulating hormone (TSH) at Baseline and every 4 weeks of treatment period and Week 28 of follow up period. Data for participants with values outside the marked reference range are reported.
Time Frame: Up to Week 28
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Participants
  Reticulocyte, maximum post Baseline: number analyzed (Participants) | 288 | 293
  Reticulocyte, maximum post Baseline | 8 | 6
  Reticulocyte Count, Absolute,maximum post Baseline: number analyzed (Participants) | 288 | 293
  Reticulocyte Count, Absolute,maximum post Baseline | 17 | 8
  White Blood Cells, maximum post Baseline: number analyzed (Participants) | 289 | 293
  White Blood Cells, maximum post Baseline | 1 | 1
  Lymphocytes, maximum post Baseline: number analyzed (Participants) | 287 | 292
  Lymphocytes, maximum post Baseline | 1 | 0
  Lymphocytes,Absolute, maximum post Baseline: number analyzed (Participants) | 287 | 292
  Lymphocytes,Absolute, maximum post Baseline | 0 | 1
  Eosinophils, maximum post Baseline: number analyzed (Participants) | 287 | 292
  Eosinophils, maximum post Baseline | 29 | 39
  Eosinophils, Absolute, maximum post Baseline: number analyzed (Participants) | 287 | 292
  Eosinophils, Absolute, maximum post Baseline | 12 | 20
  Bilirubin Total, maximum post Baseline: number analyzed (Participants) | 289 | 293
  Bilirubin Total, maximum post Baseline | 0 | 3
  ALP, maximum post Baseline: number analyzed (Participants) | 289 | 294
  ALP, maximum post Baseline | 1 | 1
  AST, maximum post Baseline: number analyzed (Participants) | 289 | 294
  AST, maximum post Baseline | 6 | 6
  ALT, maximum post Baseline: number analyzed (Participants) | 289 | 294
  ALT, maximum post Baseline | 7 | 11
  LDH, maximum post Baseline: number analyzed (Participants) | 287 | 293
  LDH, maximum post Baseline | 0 | 1
  CPK, maximum post Baseline: number analyzed (Participants) | 288 | 294
  CPK, maximum post Baseline | 28 | 27
  Cholesterol, Total, maximum post Baseline: number analyzed (Participants) | 275 | 278
  Cholesterol, Total, maximum post Baseline | 17 | 4
  Triglyceride, maximum post Baseline: number analyzed (Participants) | 275 | 278
  Triglyceride, maximum post Baseline | 16 | 2
  Glucose, maximum post Baseline: number analyzed (Participants) | 277 | 280
  Glucose, maximum post Baseline | 5 | 4
  Potassium, maximum post Baseline: number analyzed (Participants) | 288 | 294
  Potassium, maximum post Baseline | 1 | 0
  Calcium, maximum post Baseline: number analyzed (Participants) | 288 | 294
  Calcium, maximum post Baseline | 0 | 1
  Creatinine, maximum post Baseline: number analyzed (Participants) | 288 | 294
  Creatinine, maximum post Baseline | 1 | 1
  BUN, maximum post Baseline: number analyzed (Participants) | 288 | 294
  BUN, maximum post Baseline | 1 | 0
  Free T4 - Thyroxine, maximum post Baseline: number analyzed (Participants) | 289 | 294
  Free T4 - Thyroxine, maximum post Baseline | 1 | 3
  TSH, maximum post Baseline: number analyzed (Participants) | 289 | 294
  TSH, maximum post Baseline | 6 | 10
  LDL Calculated, maximum post Baseline: number analyzed (Participants) | 274 | 278
  LDL Calculated, maximum post Baseline | 102 | 62

10. Secondary Outcome: Number of Participants Referred or Not Referred to a Psychiatrist as Per Brief Summary Inventory (BSI) 53 Questionnaire up to 24 Weeks
Description: The BSI is a 53 item self-report scale used to measure nine primary symptom dimensions (somatization, obsessive-compulsive behavior, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism). Respondents rank each feeling item (e.g., "your feelings being easily hurt") on a 5-point scale where, 0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, 4=extremely (0 indicates best outcome and 4 indicates worst outcome). The total score ranged from 0 (best outcome) to 212 (worse outcome). Participants with an increase above Baseline of 25% or more on any domain subscore in BSI-53, or with an increase above Baseline of >=2 points or a score >=3 on any BSI-53 item that reflects depression, suicidality, psychotic symptoms, and hostility/aggression, were to be referred to a psychiatrist within 2 weeks.
Time Frame: Up to Week 24
Population: Safety population. Only those participants meeting the criteria of referring to psychiatrist were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Participants
  Week 4, Referred to a Psychiatrist: number analyzed (Participants) | 61 | 58
  Week 4, Referred to a Psychiatrist | 47 | 34
  Week 4, Not Referred to a Psychiatrist: number analyzed (Participants) | 61 | 58
  Week 4, Not Referred to a Psychiatrist | 14 | 24
  Week 8, Referred to a Psychiatrist: number analyzed (Participants) | 42 | 25
  Week 8, Referred to a Psychiatrist | 19 | 10
  Week 8, Not Referred to a Psychiatrist: number analyzed (Participants) | 42 | 25
  Week 8, Not Referred to a Psychiatrist | 23 | 15
  Week 12, Referred to a Psychiatrist: number analyzed (Participants) | 31 | 21
  Week 12, Referred to a Psychiatrist | 10 | 9
  Week 12, Not Referred to a Psychiatrist: number analyzed (Participants) | 31 | 21
  Week 12, Not Referred to a Psychiatrist | 21 | 12
  Week 16, Referred to a Psychiatrist: number analyzed (Participants) | 22 | 13
  Week 16, Referred to a Psychiatrist | 11 | 4
  Week 16, Not Referred to a Psychiatrist: number analyzed (Participants) | 22 | 13
  Week 16, Not Referred to a Psychiatrist | 11 | 9
  Week 20, Referred to a Psychiatrist: number analyzed (Participants) | 16 | 7
  Week 20, Referred to a Psychiatrist | 6 | 1
  Week 20, Not Referred to a Psychiatrist: number analyzed (Participants) | 16 | 7
  Week 20, Not Referred to a Psychiatrist | 10 | 6
  Week 24, Referred to a Psychiatrist: number analyzed (Participants) | 35 | 39
  Week 24, Referred to a Psychiatrist | 10 | 9
  Week 24, Not Referred to a Psychiatrist: number analyzed (Participants) | 35 | 39
  Week 24, Not Referred to a Psychiatrist | 25 | 30
  Week 28, Referred to a Psychiatrist: number analyzed (Participants) | 10 | 17
  Week 28, Referred to a Psychiatrist | 2 | 1
  Week 28, Not Referred to a Psychiatrist: number analyzed (Participants) | 10 | 17
  Week 28, Not Referred to a Psychiatrist | 8 | 16

11. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9) Score Over 28 Weeks
Description: The PHQ-9 was a standardized tests of mood/depression. This was a nine item measure with a response for each item between 0-3 where, 0=not at all, 1= several days, 2= more than half the days, 3= nearly every day. Total scores on this measure range from 0-27, with 0 being a minimum indicating no depressive symptoms, and 27 being the maximum number and severity of depressive symptoms. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-baseline values.
Time Frame: Baseline (Week 0) and Week 4, 8, 12, 16, 20, 24, 28
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Score on scale
  Week 4: number analyzed (Participants) | 265 | 274
  Week 4 | -0.3 (2.23) | -0.2 (2.32)
  Week 8: number analyzed (Participants) | 252 | 236
  Week 8 | -0.6 (2.35) | -0.6 (2.18)
  Week 12: number analyzed (Participants) | 226 | 173
  Week 12 | -0.9 (2.27) | -0.9 (2.39)
  Week 16: number analyzed (Participants) | 188 | 141
  Week 16 | -0.9 (2.25) | -0.9 (2.79)
  Week 20: number analyzed (Participants) | 167 | 130
  Week 20 | -1.0 (2.38) | -1.2 (2.66)
  Week 24: number analyzed (Participants) | 258 | 266
  Week 24 | -0.8 (2.56) | -0.6 (2.59)
  Week 28: number analyzed (Participants) | 79 | 85
  Week 28 | -0.6 (2.65) | -0.6 (2.03)

12. Secondary Outcome: Number of Participants Meeting the Referral Criteria of Psychiatric Evaluation Over 28 Weeks
Description: Participants meeting any of the following criteria were to be referred for specialist psychiatric evaluation within 2 weeks: PHQ-9 Score >=15, Two Subsequent Scores of >=10 and PHQ-9 Question 9 >=1. The PHQ -9 was a standardized tests of mood/depression. This was a nine item measure with a response for each item between 0-3 where, 0=not at all, 1= several days, 2= more than half the days, 3= nearly everyday. Total scores on this measure range from 0-27, with 0 being a minimum indicating no depressive symptoms, and 27 being the maximum number and severity of depressive symptoms. Only categories with data available at the indicated time points have been presented. Categories with null values for all the arms have not been presented.
Time Frame: Up to 28 Weeks
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Participants
  Week 4, PHQ-9 Score >=15: number analyzed (Participants) | 273 | 278
  Week 4, PHQ-9 Score >=15 | 2 | 0
  Week 4, Two Subsequent Scores of >=10: number analyzed (Participants) | 273 | 278
  Week 4, Two Subsequent Scores of >=10 | 3 | 2
  Week 4, PHQ-9 Question 9 >=1: number analyzed (Participants) | 273 | 278
  Week 4, PHQ-9 Question 9 >=1 | 3 | 3
  Week 4, Referred to a Psychiatrist: number analyzed (Participants) | 273 | 278
  Week 4, Referred to a Psychiatrist | 3 | 2
  Week 4, Not Referred to a Psychiatrist: number analyzed (Participants) | 273 | 278
  Week 4, Not Referred to a Psychiatrist | 1 | 2
  Week 8, Two Subsequent Scores of >=10: number analyzed (Participants) | 252 | 241
  Week 8, Two Subsequent Scores of >=10 | 1 | 2
  Week 8, PHQ-9 Question 9 >=1: number analyzed (Participants) | 252 | 241
  Week 8, PHQ-9 Question 9 >=1 | 4 | 1
  Week 8, Referred to a Psychiatrist: number analyzed (Participants) | 252 | 241
  Week 8, Referred to a Psychiatrist | 1 | 1
  Week 8, Not Referred to a Psychiatrist: number analyzed (Participants) | 252 | 241
  Week 8, Not Referred to a Psychiatrist | 3 | 1
  Week 12, Two Subsequent Scores of >=10: number analyzed (Participants) | 228 | 177
  Week 12, Two Subsequent Scores of >=10 | 0 | 1
  Week 12, PHQ-9 Question 9 >=1: number analyzed (Participants) | 228 | 177
  Week 12, PHQ-9 Question 9 >=1 | 2 | 0
  Week 12, Not Referred to a Psychiatrist: number analyzed (Participants) | 228 | 177
  Week 12, Not Referred to a Psychiatrist | 2 | 1
  Week 16, PHQ-9 Score >=15: number analyzed (Participants) | 190 | 144
  Week 16, PHQ-9 Score >=15 | 1 | 0
  Week 16, PHQ-9 Question 9 >=1: number analyzed (Participants) | 190 | 144
  Week 16, PHQ-9 Question 9 >=1 | 2 | 0
  Week 16, Not Referred to a Psychiatrist: number analyzed (Participants) | 190 | 144
  Week 16, Not Referred to a Psychiatrist | 2 | 0
  Week 20, PHQ-9 Question 9 >=1: number analyzed (Participants) | 168 | 131
  Week 20, PHQ-9 Question 9 >=1 | 1 | 0
  Week 20, Not Referred to a Psychiatrist: number analyzed (Participants) | 168 | 131
  Week 20, Not Referred to a Psychiatrist | 1 | 0
  Week 24, PHQ-9 Score >=15: number analyzed (Participants) | 262 | 270
  Week 24, PHQ-9 Score >=15 | 1 | 0
  Week 24, Two Subsequent Scores of >=10: number analyzed (Participants) | 262 | 270
  Week 24, Two Subsequent Scores of >=10 | 0 | 1
  Week 24, PHQ-9 Question 9 >=1: number analyzed (Participants) | 262 | 270
  Week 24, PHQ-9 Question 9 >=1 | 1 | 2
  Week 24, Not Referred to a Psychiatrist: number analyzed (Participants) | 262 | 270
  Week 24, Not Referred to a Psychiatrist | 2 | 2
  Week 28, PHQ-9 Score >=15: number analyzed (Participants) | 79 | 86
  Week 28, PHQ-9 Score >=15 | 2 | 0
  Week 28, Two Subsequent Scores of >=10: number analyzed (Participants) | 79 | 86
  Week 28, Two Subsequent Scores of >=10 | 2 | 0
  Week 28, PHQ-9 Question 9 >=1: number analyzed (Participants) | 79 | 86
  Week 28, PHQ-9 Question 9 >=1 | 2 | 0
  Week 28, Not Referred to a Psychiatrist: number analyzed (Participants) | 79 | 86
  Week 28, Not Referred to a Psychiatrist | 3 | 0

13. Secondary Outcome: Change From Baseline in Hearing Handicap Inventory for the Elderly-Screening (HHIE-S) Over 24 Weeks
Description: HHIE-S assessed participants by handicap category: no handicap (0 to 8 points); mild/moderate handicap (10 to 24 points); severe handicap (26-40 points). Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-baseline values.
Time Frame: Baseline (Week 0) and Week 4, 8, 12, 16, 20, 24
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Score on scale
  Week 4: number analyzed (Participants) | 83 | 88
  Week 4 | -0.0 (0.96) | -0.2 (0.86)
  Week 8: number analyzed (Participants) | 77 | 74
  Week 8 | -0.1 (1.14) | -0.1 (0.69)
  Week 12: number analyzed (Participants) | 70 | 55
  Week 12 | -0.2 (1.01) | -0.1 (0.52)
  Week 16: number analyzed (Participants) | 58 | 39
  Week 16 | -0.1 (0.79) | -0.1 (0.32)
  Week 20: number analyzed (Participants) | 51 | 35
  Week 20 | -0.2 (0.78) | -0.1 (0.34)
  Week 24: number analyzed (Participants) | 79 | 81
  Week 24 | -0.2 (1.02) | -0.2 (1.10)

14. Secondary Outcome: Change From Baseline in Dizziness Handicap Inventory (DHI) Over 24 Weeks
Description: DHI assessed participants by handicap category: no handicap (0 to 14 points); mild handicap (16 to 34 points); moderate handicap (36 to 52 points); severe handicap (54 points). Increase from Baseline of <6 points, 6 to <12 points and 12 points. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-baseline values.
Time Frame: Baseline (Week 0) and Week 4, 8, 12, 16, 20, 24
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Score on scale
  Week 4: number analyzed (Participants) | 82 | 86
  Week 4 | -0.3 (2.65) | 0.3 (1.26)
  Week 8: number analyzed (Participants) | 74 | 74
  Week 8 | -0.5 (2.68) | -0.1 (1.02)
  Week 12: number analyzed (Participants) | 70 | 54
  Week 12 | -0.2 (3.78) | -0.1 (0.38)
  Week 16: number analyzed (Participants) | 57 | 38
  Week 16 | 0.1 (1.38) | -0.1 (1.18)
  Week 20: number analyzed (Participants) | 49 | 35
  Week 20 | 0.2 (2.34) | -0.1 (1.24)
  Week 24: number analyzed (Participants) | 78 | 78
  Week 24 | 0.7 (5.72) | 0.2 (2.41)

15. Secondary Outcome: Number of Participants Responding to Tinnitus Ototoxicity Monitoring Interview (TOMI) Questionnaire Over 24 Weeks
Description: Participants who developed tinnitus were monitored by use of the TOMI. The numbers of participants with pre-existing tinnitus, new tinnitus, increased/decreased loudness of tinnitus, or increased/decreased duration of tinnitus, pulsing quality of tinnitus were assessed.
Time Frame: Up to Week 24
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Participants
  Persistent TInnitus since treatment, yes: number analyzed (Participants) | 131 | 114
  Persistent TInnitus since treatment, yes | 16 | 5
  Type of Tinnitus, Ringing: number analyzed (Participants) | 15 | 5
  Type of Tinnitus, Ringing | 11 | 2
  Type of Tinnitus, Buzzing: number analyzed (Participants) | 15 | 5
  Type of Tinnitus, Buzzing | 3 | 0
  Type of Tinnitus, Hissing: number analyzed (Participants) | 15 | 5
  Type of Tinnitus, Hissing | 1 | 0
  Type of Tinnitus, Whistle: number analyzed (Participants) | 15 | 5
  Type of Tinnitus, Whistle | 1 | 1
  Type of Tinnitus, Hum: number analyzed (Participants) | 15 | 5
  Type of Tinnitus, Hum | 3 | 0
  Type of Tinnitus, Other: number analyzed (Participants) | 15 | 5
  Type of Tinnitus, Other | 0 | 2
  Tinnitus - Pulsing Quality, Yes: number analyzed (Participants) | 15 | 5
  Tinnitus - Pulsing Quality, Yes | 3 | 0
  Tinnitus Location, Left Ear only: number analyzed (Participants) | 15 | 5
  Tinnitus Location, Left Ear only | 2 | 0
  Tinnitus Location, Right Ear only: number analyzed (Participants) | 15 | 5
  Tinnitus Location, Right Ear only | 4 | 1
  Tinnitus Location, Both ears: number analyzed (Participants) | 15 | 5
  Tinnitus Location, Both ears | 7 | 1
  Tinnitus Location, Inside head: number analyzed (Participants) | 15 | 5
  Tinnitus Location, Inside head | 2 | 2
  Tinnitus Location, Other: number analyzed (Participants) | 15 | 5
  Tinnitus Location, Other | 0 | 1
  Tinnitus Louder on right side of head: number analyzed (Participants) | 14 | 4
  Tinnitus Louder on right side of head | 5 | 1
  Tinnitus Louder on left side of head: number analyzed (Participants) | 14 | 4
  Tinnitus Louder on left side of head | 2 | 0
  Tinnitus Equal on both side of head: number analyzed (Participants) | 14 | 4
  Tinnitus Equal on both side of head | 7 | 3
  Slightly loud tinnitus: number analyzed (Participants) | 16 | 4
  Slightly loud tinnitus | 3 | 0
  Moderately loud tinnitus: number analyzed (Participants) | 16 | 4
  Moderately loud tinnitus | 6 | 1
  How much of Time Tinnitus Present, Occasionally: number analyzed (Participants) | 15 | 4
  How much of Time Tinnitus Present, Occasionally | 4 | 3
  How much of Time Tinnitus Present,Some of the Time: number analyzed (Participants) | 15 | 4
  How much of Time Tinnitus Present,Some of the Time | 3 | 0
  How much of Time Tinnitus Present,Most of the Time: number analyzed (Participants) | 15 | 4
  How much of Time Tinnitus Present,Most of the Time | 5 | 0
  How much of Time Tinnitus Present,Always: number analyzed (Participants) | 15 | 4
  How much of Time Tinnitus Present,Always | 3 | 1
  How much of a Problem is Tinnitus, Slight: number analyzed (Participants) | 16 | 4
  How much of a Problem is Tinnitus, Slight | 5 | 1
  How much of a Problem is Tinnitus, Moderate: number analyzed (Participants) | 16 | 4
  How much of a Problem is Tinnitus, Moderate | 2 | 0
  How much of a Problem is Tinnitus, Big: number analyzed (Participants) | 16 | 4
  How much of a Problem is Tinnitus, Big | 1 | 0
  Has the Sound of Tinnitus Changed, Yes: number analyzed (Participants) | 15 | 4
  Has the Sound of Tinnitus Changed, Yes | 1 | 0
  Has Loudness of Tinnitus Changed,Yes,Louder Now: number analyzed (Participants) | 15 | 4
  Has Loudness of Tinnitus Changed,Yes,Louder Now | 1 | 0
  Has Loudness of Tinnitus Changed,Yes,Quieter Now: number analyzed (Participants) | 15 | 4
  Has Loudness of Tinnitus Changed,Yes,Quieter Now | 1 | 0
  Amount of TimeTinnitus PresentChanged,Yesmoreoften: number analyzed (Participants) | 15 | 4
  Amount of TimeTinnitus PresentChanged,Yesmoreoften | 1 | 0
  Amount of TimeTinnitus PresentChanged,Yeslessoften: number analyzed (Participants) | 15 | 4
  Amount of TimeTinnitus PresentChanged,Yeslessoften | 1 | 1

16. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) by Dual Energy X-ray Absorptiometry (DXA) Over 72 Weeks
Description: Bone mineral density scans of the left proximal femur (total hip) and anterior-posterior lumbar spine were obtained by use of DXA, at Baseline, at end of therapy, and 1 year (48 weeks) after end of therapy. In case of abnormality or surgery of the left hip, the right hip was to be used. If both hips were affected, the participant was not eligible for DXA. Vertebrae L1 to L4 had to be completely scanned. At least 3 vertebrae had to be free of any abnormalities potentially interfering with DXA analysis (eg, fractures, large osteophytes), otherwise the participant was not eligible for DXA. Baseline was defined at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-baseline values. Percentage change from Baseline = (change from Baseline / Baseline value) * 100. Least square means and 95% confidence interval has been presented.
Time Frame: Baseline (Week 0) and Week 72
Population: Safety Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 296 | 298
Percent change
  Lumbar Spine BMD: number analyzed (Participants) | 182 | 164
  Lumbar Spine BMD | 0.385 [-0.403 to 1.173] | -0.104 [-0.827 to 0.618]
  Femur BMD: number analyzed (Participants) | 179 | 158
  Femur BMD | 0.435 [-0.196 to 1.065] | -0.063 [-0.644 to 0.519]
Statistical Analysis 1: Comparison: Alitretinoin 30 mg vs Placebo; Lumbar Spine BMD; Test type: Superiority; p = 0.179, ANCOVA — The analysis of covariance model includes treatment, age at Baseline, gender, menopausal status of females, baseline BMD score and duration of treatment exposure (<12weeks, >=12 weeks) as covariates; Mean Difference (Net) = 0.489, 95% CI 2-sided [-0.226 to 1.204]
Statistical Analysis 2: Comparison: Alitretinoin 30 mg vs Placebo; Femur BMD; Test type: Superiority; p = 0.089, ANCOVA — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Net) = 0.497, 95% CI 2-sided [-0.077 to 1.071]

17. Secondary Outcome: Number of Participants With Adequecy of Images Assessed by X-ray Evaluation of Bones
Description: X-ray evaluations was done at Baseline (Week 0), end of therapy and at follow up period (Week 72). X-ray evaluations was done for Lateral C-Spine, Lateral T-Spine and Calcaneous. The images were evaluated as optimal, readable (but not optimal) or not readable.
Time Frame: Up to Week 72
Population: Safety Population. Only those participants who had X-ray evaluations were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 244 | 243
Participants
  Baseline,Lateral C-Spine, Optimal | 73 | 85
  Baseline,Lateral C-Spine,Readable | 171 | 158
  Baseline,Lateral T-Spine,Readable | 229 | 234
  Baseline,Lateral T-Spine,Not Readable | 15 | 9
  Baseline, Calcaneous, Optimal | 195 | 191
  Baseline, Calcaneous, Readable | 48 | 51
  Baseline, Calcaneous, Not Readable | 1 | 1
  End of Therapy,Lateral C-Spine,Optimal | 80 | 87
  End of Therapy,Lateral C-Spine,Readable | 162 | 146
  End of Therapy,Lateral C-Spine, Not Readable | 2 | 10
  End of Therapy, Lateral T-Spine, Readable | 232 | 229
  End of Therapy, Lateral T-Spine, Not Readable | 12 | 14
  End of Therapy, Calcaneous, Optimal | 196 | 182
  End of Therapy, Calcaneous, Readable | 40 | 44
  End of Therapy, Calcaneous, Not Readable | 8 | 17
  Week 72, Lateral C-Spine, Optimal | 39 | 38
  Week 72, Lateral C-Spine, Readable | 151 | 134
  Week 72, Lateral C-Spine, Not Readable | 0 | 1
  Week 72, Lateral C-Spine, Missing | 54 | 70
  Week 72, Lateral T-Spine, Readable | 183 | 168
  Week 72, Lateral T-Spine, Not Readable | 7 | 5
  Week 72, Lateral T-Spine, Missing | 54 | 70
  Week 72, Calcaneous, Optimal | 141 | 119
  Week 72, Calcaneous, Not Readable | 6 | 4
  Week 72, Calcaneous, Missing | 54 | 70
  Week 72, Calcaneous, Readable | 43 | 50

18. Secondary Outcome: Number of Participants With Adverse Ophthalmological Change as Assessed by Fundus Photography - Intraocular Pressure
Description: An adverse change was defined as a change from normal at Baseline to abnormal at end of therapy, or as a worsening from Baseline for either or both eyes. A missing adverse change was defined as missing results at Baseline and end of therapy, or missing result at Baseline and abnormal at end of therapy, or normal at Baseline and missing result at end of therapy, or abnormal at Baseline and missing result at end of therapy, for both eyes or one eye when the other eye was not concerned by an adverse change. Other changes from Baseline to end of therapy was considered as no adverse change. Optic disc, macula, and retinal periphery were assessed by fundoscopy after pupil dilation using tropicamide.
Time Frame: Up to Week 24
Population: Safety Population. Only those participants who had ophthalmological evaluations were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 180 | 186
Participants
  Participants with an Adverse Change, No | 152 | 146
  Participants with an Adverse Change, Yes | 0 | 1
  Participants with an Adverse Change, Missing | 28 | 39
  Baseline, Normal | 177 | 183
  Baseline, Abnormal | 3 | 1
  Baseline, Missing | 0 | 2
  End of Therapy, Normal | 152 | 146
  End of Therapy, Abnormal | 1 | 1
  End of Therapy, Missing | 27 | 39
  Worsened from Baseline, No: number analyzed (Participants) | 3 | 1
  Worsened from Baseline, No | 2 | 1
  Worsened from Baseline, Missing: number analyzed (Participants) | 3 | 1
  Worsened from Baseline, Missing | 1 | 0

19. Secondary Outcome: Number of Participants With Adverse Audiological Change as Assessed by Puretone Audiogram at Highest Frequency
Description: An adverse change was defined as a change from normal at Baseline to abnormal at end of therapy. A missing adverse change was defined as missing results at Baseline and end of therapy, or missing result at Baseline and abnormal at end of therapy, or normal at Baseline and missing result at end of therapy. Other changes from Baseline to end of therapy are considered as no adverse change. All puretone testing used a modified Hughson-Westlake procedure with 5 decibel (dB) step size.
Time Frame: Up to Week 24
Population: Safety Population. Only those participants who had audiologic evaluations were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Alitretinoin 30 mg | Placebo
Number analyzed (Participants) | 149 | 147
Participants
  Participants with adverse change, No | 131 | 125
  Participants with adverse change, Yes | 4 | 10
  Participants with adverse change, Missing | 14 | 12
  Baseline, Normal | 57 | 69
  Baseline, Abnormal | 91 | 75
  Baseline, Missing | 1 | 3
  End of Therapy, Normal | 48 | 55
  End of Therapy, Abnormal | 75 | 71
  End of Therapy, Missing | 26 | 21

ADVERSE EVENTS:
Time Frame: AEs were collected up to follow up period (up to Week 28). Treatment emergent SAEs and nSAEs (up to Week 24) has been presented.
Description: Safety Population was used for the analysis of safety data.
Arm/Group | Alitretinoin 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/296 | 2/298
Serious Adverse Events (participants affected / at risk) | 7/296 | 3/298
Other Adverse Events (participants affected / at risk) | 108/296 | 36/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alitretinoin 30 mg (N=296) | Placebo (N=298)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Granuloma (General disorders) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
ACCIDENT AT HOME (Injury, poisoning and procedural complications) | 0 | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 1
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alitretinoin 30 mg (N=296) | Placebo (N=298)
Upper respiratory tract infection (Infections and infestations) | 20 | 13
Headache (Nervous system disorders) | 87 | 24
Flushing (Vascular disorders) | 17 | 1
Nausea (Gastrointestinal disorders) | 22 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.